CLINICAL TRIAL: NCT00422188
Title: Phase 1, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Sequential Dose-Escalation Study of the Pharmacokinetics, Safety, and Efficacy of ATX-101 (Sodium Deoxycholate for Injection) Intralipomal Injections for the Treatment of Superficial Lipomas
Brief Title: Deoxycholic Acid Injection for the Treatment of Superficial Lipomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATX-101-06-04
Record Dates: First submitted 2007-01-11; First posted 2007-01-15 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Lipoma
MeSH Terms: conditions — Lipoma | interventions — Deoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Deoxycholic Acid Injection 0.5% (Experimental): Participants received 0.5% deoxycholic acid administered at a volume dependent on the size of the lipoma up to a maximum of 5 mL for 2 treatments at 28-day intervals.
  Interventions: Drug: Deoxycholic Acid Injection
- Deoxycholic Acid Injection 1.0% (Experimental): Participants received 1.0% deoxycholic acid administered at a volume dependent on the size of the lipoma up to a maximum of 5 mL for 2 treatments at 28-day intervals.
  Interventions: Drug: Deoxycholic Acid Injection
- Deoxycholic Acid Injection 2.0% (Experimental): Participants received 2.0% deoxycholic acid administered at a volume dependent on the size of the lipoma up to a maximum of 5 mL for 2 treatments at 28-day intervals.
  Interventions: Drug: Deoxycholic Acid Injection
- Deoxycholic Acid Injection 4.0% (Experimental): Participants received 4.0% deoxycholic acid administered at a volume dependent on the size of the lipoma up to a maximum of 5 mL for 2 treatments at 28-day intervals.
  Interventions: Drug: Deoxycholic Acid Injection
- Placebo (Placebo Comparator): Participants received matching vehicle placebo administered at a volume dependent on the size of the lipoma up to a maximum of 5 mL for 2 treatments at 28-day intervals.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deoxycholic Acid Injection — Administered via intralipomal injection.
  Other Names: ATX-101; Sodium deoxycholate
  Arms: Deoxycholic Acid Injection 0.5%; Deoxycholic Acid Injection 1.0%; Deoxycholic Acid Injection 2.0%; Deoxycholic Acid Injection 4.0%
Drug: Placebo — Administered via intralipomal injection.
  Arms: Placebo

SUMMARY:
The purpose of this research is to compare the safety and effectiveness of 4 different concentrations of deoxycholic acid injection against a placebo in the treatment of superficial lipomas.

DETAILED DESCRIPTION:
A lipoma is a fatty lump typically located on the trunk, shoulder, arms or legs. For the purposes of this study, only lipomas on the trunk, arms, legs, or neck were treated. (Lipomas on the face, wrists, hands, lower portion of the spine, genitals, ankles, or feet were not treated.)

ELIGIBILITY:
Inclusion Criteria:

* One or more lipomas, based on clinical diagnosis, which are accessible for treatment and assessment, are quantifiable along at least 2 perpendicular diameters, and have the following characteristics:

  * History of slow growth followed by dormancy, and stable for at least 6 months.
  * Greatest length by greatest perpendicular width between 1 and 16 square centimeters, inclusive
  * Discrete, oval to rounded in shape, not hard or attached to underlying tissue
  * Located on the trunk, arms, legs, or neck
* Stable body weight with a body mass index of less than 30 kg/m²
* Signed informed consent

Exclusion Criteria:

* Absence of significant medical conditions that could affect safety
* History of surgical treatment for lipomas
* Treatment with an investigational agent within 30 days before ATX-101 treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Assessments of Safety with Laboratory tests | up to 16 weeks
Assessments of Safety with ECG | up to 16 weeks
Assessments of Safety with Medical Evaluations | up to 16 weeks

SECONDARY OUTCOMES:
Lipoma size reduction | up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stacy R. Smith, M.D., Principal Investigator — Therapeutics Clinical Research
Locations (1):
- Therapeutics Clinical Research, San Diego, California, United States